CLINICAL TRIAL: NCT02776579
Title: Girls in the Weight Room: Assessing the Influence of a Female School-based Strength & Conditioning Specialist on the Health of High School Girls
Brief Title: Effect of a Female Strength & Conditioning Specialist on High School Girls' Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Grant Park
Record Dates: First submitted 2016-05-09; First posted 2016-05-18 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Physical Inactivity; Low Physical Fitness
Keywords: Resistance Training; Muscle Strength
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Girls-only resistance training (Experimental): 8 weeks of 2-3x/week girls-only resistance training class with a female strength and conditioning specialist.
  Interventions: Other: Girls-only resistance training
- No resistance training (No Intervention): 8 weeks of usual activity.

INTERVENTIONS:
Other: Girls-only resistance training
  Arms: Girls-only resistance training

SUMMARY:
The majority of today's youth do not engage in enough physical activity (PA) to maintain good health. Low PA levels are associated with poor health (e.g. diabetes, high blood pressure) and early mortality. Girls are less likely than boys to be active, and their rates of participation drop off more steeply during adolescence. Girls report many barriers to exercise, including transportation issues and feeling self-conscious about their appearance and abilities. School-based PA programs that try to improve health, mainly through aerobic exercise and education, have had a small effect to date. However, the few programs that included resistance training as the focus showed strong improvements in health related measures. In this project, we will examine the effect of a female strength and conditioning specialist on decreasing barriers and increasing the overall health of high school girls, with the delivery of in-school, girls-only resistance training programs. We will see if physical and mental health changes with the training, and how the presence of the S & C specialist affects the girls' social interactions within the school. The results will help individuals in the education sector plan programs and services to improve overall youth and school health.

ELIGIBILITY:
Inclusion Criteria:

* Grades 7 to 12 at Grant Park High School
* do not participate on organized sports teams
* self-report as not meeting the recommended amount of 60 min of Moderate-Vigorous Physical Activity per day

Exclusion Criteria:

* engaged in regular resistance training activities within the previous 6 months
* health condition or injury that would put them at risk during testing/training

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
1 Repetition Maximum leg press | Change from Baseline and at 8 weeks

SECONDARY OUTCOMES:
1 Repetition Maximum bench press | Baseline and at 8 weeks
Grip strength dynamometry | Baseline and at 8 weeks
  The average of three repetitions for each hand will be used in analysis
mCAFT for aerobic fitness | Baseline and at 8 weeks
Physical activity levels | Baseline and at 8 weeks
  Average daily minutes spent in Sedentary, Low, Moderate and Vigorous intensity activity over 5 days will be measured via an accelerometer worn around the waist.
Physical Self-Perception Profile | Baseline and at 8 weeks
  36 item questionnaire; scores for embedded scales of "Strength Competence", "Physical Self-Worth", "Global Self-Worth", and "Attractive Body Adequacy" will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Parsons, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No